CLINICAL TRIAL: NCT04985357
Title: Defining the Clinical Potential of Mass Response As a Biomarker for Patient Tumor Sensitivity to Drugs
Status: Withdrawn | Type: Observational
Why Stopped: Abandoned prior to launch.
Sponsor: Travera Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: TRV-002
Record Dates: First submitted 2021-07-15; First posted 2021-08-02 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Stage III Breast Cancer; Stage IV Breast Cancer; Stage III Lung Cancer; Stage IV Lung Cancer; AML; Multiple Myeloma in Relapse; Carcinoma; Carcinoma, Pancreatic; Carcinoma of Lung; Carcinoma, Non-Small-Cell Lung; Carcinoma Breast; Carcinoma Prostate; Carcinoma, Hepatocellular; Carcinoma, Renal Cell; Carcinoma, Neuroendocrine; Carcinoma, Small Cell Lung; Carcinoma, Ovarian; Carcinoma Bladder; Carcinoma of Esophagus; Carcinoma Cervix; Carcinoma, Thymic; Carcinoma, Ductal; Carcinoma of the Head and Neck; Carcinoma of the Lip; Carcinoma of the Oral Cavity; Carcinoma of Unknown Primary; Carcinoma of the Skin; Carcinoma of the Anus; Carcinoma of the Larynx; Carcinoma of the Penis; Carcinoma of the Oropharynx; Carcinoma of the Appendix; Carcinoma of the Paranasal Sinus; Carcinoma of the Vulva; Malignant Pleural Effusion; Malignant Ascites; Mesothelioma; Cholangiocarcinoma
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms; Carcinoma; Pancreatic Neoplasms; Carcinoma, Non-Small-Cell Lung; Prostatic Neoplasms; Carcinoma, Hepatocellular; Carcinoma, Renal Cell; Carcinoma, Neuroendocrine; Small Cell Lung Carcinoma; Ovarian Neoplasms; Urinary Bladder Neoplasms; Esophageal Neoplasms; Uterine Cervical Neoplasms; Thymoma; Carcinoma, Ductal; Lip Neoplasms; Mouth Neoplasms; Neoplasms, Unknown Primary; Anus Neoplasms; Laryngeal Neoplasms; Penile Neoplasms; Oropharyngeal Neoplasms; Appendiceal Neoplasms; Paranasal Sinus Neoplasms; Vulvar Neoplasms; Pleural Effusion, Malignant; Mesothelioma; Cholangiocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (6):
- Carcinoma-Associated Malignant Fluid: Diagnosis of any kind of carcinoma with a malignant fluid (pleural effusion or ascites) where drainage is clinically indicated as part of SOC, and a new course of treatment is upcoming.
- Carcinoma Solid Tissue Specimen: Diagnosis of any kind of carcinoma where a needle biopsy or tissue resection is clinically indicated as part of SOC, and a new course of treatment is upcoming.
- Multiple Myeloma: Diagnosis of relapsed multiple myeloma where bone marrow biopsy is clinically indicated as part of SOC, and a new course of treatment is upcoming.
- Acute myelogenous leukemia (AML): Diagnosis of acute myelogenous leukemia where a blood draw or bone marrow biopsy is clinically indicated as part of SOC, and a new course of treatment is upcoming.
- Triple Negative Breast Cancer (TNBC): Diagnosis of Stage IV Triple Negative Breast Cancer where a needle biopsy is clinically indicated as part of SOC, and a new course of treatment is upcoming.
- Peripheral Blood Cell Immune Competency: Diagnosis of any cancer where a blood draw is clinically indicated as part of SOC, a new course of treatment is upcoming, and checkpoint inhibitor therapy being considered for next line of treatment.

SUMMARY:
The primary objective of this study, sponsored by Travera in Massachusetts, is to validate whether the mass response biomarker has potential to predict response of patients to specific therapies or therapeutic combinations using isolated tumor cells from varying cancers and biopsy formats.

ELIGIBILITY:
Inclusion Criteria:

* Sample collection or biopsy of tumor is clinically indicated as part of SOC
* Prior to preceding onto therapy for treatment

Exclusion Criteria:

* Unable to obtain sufficient sample

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: General population with cohort matched diagnoses.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-11 (Estimated); Primary Completion 2028-05 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Best overall response (BOR) | up to 24 months
  The best overall response to therapy over 24 months will be captured for correlation with test outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Stevens, Ph.D., Principal Investigator — Travera Inc; Robert Kimmerling, Ph.D., Principal Investigator — Travera Inc

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://www.travera.com